CLINICAL TRIAL: NCT03595384
Title: Feasibility of a Soccer-based Adaptation of the Diabetes Prevention Program
Brief Title: Soccer-based Adaptation of the Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Diabetes Translation Research (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Roberto Felipe Lobelo, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00100342; P30DK111024 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Diabetes
Keywords: Behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a longitudinal pre-post pilot intervention study evaluating feasibility of implementation of a soccer-based Diabetes Prevention Program and preliminary changes in physical activity and diet-related measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soccer-based adaptation to the DPP (Experimental): Hispanic overweight male participants taking part in a 24 week soccer program as part of diabetes prevention.
  Interventions: Behavioral: Soccer-based adaptation to the DPP

INTERVENTIONS:
Behavioral: Soccer-based adaptation to the DPP — Participants will complete online education modules during an initial 12 week conditioning phase where they will participate in soccer drills and other fitness routines (two 1-hour sessions per week). At the 12 week mark participants will transition onto a soccer league team for the following 12 weeks where they will continue to complete online modules and meet with the soccer coach monthly.
  During the soccer sessions and games participants will be fitted with a wearable soccer-specific device to measure how much they move and their heart rate. In addition, they will also be asked to wear a Garmin fitness tracker for the duration of the study to measure steps and moderate and vigorous activity.
  The online education will be a version of the Diabetes Prevention Program and can be completed on a phone or computer with internet access.

SUMMARY:
This is a longitudinal pre-post pilot intervention study evaluating feasibility of implementation of a soccer-based Diabetes Prevention Program (DPP) and preliminary changes in physical activity and diet-related measures. Overweight participants at high risk for type 2 diabetes mellitus (T2DM) will be recruited through soccer interest groups, local leagues and Hispanic health organizations. After a baseline assessment visit, participants will attend soccer practice twice a week for 12 weeks while completing the National Diabetes Prevention Program (NDPP) core curriculum online modules with facilitated discussion by trained coaches during each soccer practice. Participants will then be invited to join an established small-sided soccer league in their community (for 12 weeks) offering one game per week and will also complete the NDPP maintenance modules and physical activity and diet self-tracking via mobile health technologies. After the core (first 12 weeks) and maintenance intervention periods (second 12 weeks) baseline measurements will be repeated. Data on the feasibility of this DPP soccer-based adaptation will inform future randomized, controlled trials testing the effectiveness of this translation model to reduce T2DM risk while extrapolating to other sports-based adaptation and age, gender and racial sub-populations.

DETAILED DESCRIPTION:
The Diabetes Prevention Program (DPP) has been successful in reducing the incidence of type 2 diabetes mellitus (T2DM) through moderate weight loss and increased physical activity, and evidence from the original DPP suggests that adoption of increased physical activity (PA) habits are maintained up to 10 years among intervention participants when compared to control. Hispanic males are difficult to engage in traditional lifestyle or non-communicable chronic disease (NCDs) prevention interventions, yet, they have high rates of obesity and are at high risk for NCDs, particularly T2DM. Small-sided recreational soccer (RS) 6-12 month interventions have shown to be effective to achieve 5% weight loss and reduce cardio-metabolic risk, stemming from its varied movement patterns and highly functional training. Although proven cost-effectiveness and currently expanding in Europe, RS cardio-metabolic preventive interventions have not been tested in U.S. populations.

To fill this gap in health promotion, the goal for this proposal is to utilize the local Hispanic community's interest in soccer as a vehicle to deliver an adapted DPP among male, overweight, Latino adults at high T2DM risk. The researchers will test the following central hypothesis: A soccer-based adaptation to the DPP, can be feasibly implemented in a middle-age Latino men population at high risk for T2DM. In lieu of the traditional walking or exercise program, participants will be enrolled in 12 weeks of soccer conditioning followed by 12 weeks of small-sided soccer league play. National Diabetes Prevention Program (NDPP) online core and maintenance modules will also be facilitated by trained coaches during soccer practice for the first 12 weeks and through monthly in-person meetings the last 12 weeks. Physical activity volume, sleep and sedentary time will be tracked objectively with wearable devices linked to an innovative research smartphone app that provides data to the researchers and tailored in-app notifications and surveys to the participant. Additionally, the study will assess implementation feasibility and explore preliminary signals for improvements in objectively-measured PA, dietary behaviors, physical fitness and body composition and quality of life outcomes with the soccer-based DPP adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latino men aged 35-55 years
* Body Mass Index (BMI) ≥ 25 kg/m^2
* Centers for Disease Control and Prevention (CDC) pre-diabetes risk score ≥ 9
* Not currently engaged in soccer practice or league or other physical activity or lifestyle intervention program
* Ability to read in English or Spanish and provide inform consent

Exclusion Criteria:

* T2DM diagnosis or medication
* BMI ≥ 41
* Resting blood pressure ≥165/100 at screening
* Any mobility issues or contraindications for high intensity interval training (HIIT) physical activity program

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-04-29 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2018-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Lobelo, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Rollins School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data supporting the conclusions of this study are available for sharing with other researchers.
Time Frame: Raw data are available for sharing following publication of the results of this study.
Access Criteria: Access to the data can be obtained by emailing the study investigators.

REFERENCES:
- [Background] Frediani JK, Bienvenida AF, Li J, Higgins MK, Lobelo F. Physical fitness and activity changes after a 24-week soccer-based adaptation of the U.S diabetes prevention program intervention in Hispanic men. Prog Cardiovasc Dis. 2020 Nov-Dec;63(6):775-785. doi: 10.1016/j.pcad.2020.06.012. Epub 2020 Jun 27. PMID 32603753
- [Result] Frediani JK, Li J, Bienvenida A, Higgins MK, Lobelo F. Metabolic Changes After a 24-Week Soccer-Based Adaptation of the Diabetes Prevention Program in Hispanic Males: A One-Arm Pilot Clinical Trial. Front Sports Act Living. 2021 Nov 12;3:757815. doi: 10.3389/fspor.2021.757815. eCollection 2021. PMID 34870194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in April through July of 2018 and all follow-up was completed by December 16, 2018.
Groups:
- Soccer-based Adaptation to the Diabetes Prevention Program (DPP): Participants taking part in a 24 week soccer program as part of diabetes prevention. Participants completed online education modules during an initial 12 week conditioning phase where they participated in soccer drills and other fitness routines (two 1-hour sessions per week). At the 12 week mark participants transitioned onto a soccer league team for the following 12 weeks where they continued to complete online modules and meet with the soccer coach monthly. During the soccer sessions and games participants were fitted with a wearable soccer-specific device to measure how much they move and their heart rate. Additionally, they were asked to wear a Garmin fitness tracker for the duration of the study to measure steps and moderate and vigorous activity.
Period: Overall Study
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Started | 41
Completed Week 12 Assessment | 37
Completed (Completed Week 24 Assessment) | 25
Not Completed | 16
Not completed — Other time commitments | 8
Not completed — Changes to session time | 7
Not completed — Relocation out of country | 1

BASELINE CHARACTERISTICS:
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41
Family history of diabetes [Count of Participants; unit: Participants] — Family history of diabetes is defined as having a sibling and/or parent with diabetes.
  Participants | 21
Country of origin [Count of Participants; unit: Participants]
  Mexico | 16
  Venezuela | 4
  Ecuador | 3
  Guatemala | 4
  Colombia | 7
  Other | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 32.7 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing the Study
Description: Feasibility of the study will be assessed by the number of participants completing the study.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
Participants | 25

2. Primary Outcome: Participant Satisfaction With Overall Program
Description: Participants indicate how satisfied they were with the overall program with a single item which was scored on a scale of 1 (poor) to 10 (excellent).
Time Frame: Week 24
Population: This analysis includes participants who completed the Week 24 study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 25
units on a scale | 9.9 (0.3)

3. Secondary Outcome: Weight
Description: Body composition will be assessed by weight in kilograms (kg).
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
kilograms
  Baseline | 93.9 (2.2)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 90.7 (2.0)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 90.1 (2.0)

4. Secondary Outcome: Steps Per Day
Description: Participants will be asked to wear a Garmin fitness tracker throughout the study and physical activity will be measured as steps taken per day.
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: Steps per day
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
Steps per day
  Baseline | 12644.5 (769)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 11131.9 (807.7)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 9691.2 (993.6)

5. Secondary Outcome: Intake of Added Sugars
Description: The dietary behavior of consumption of added sugars was measured by using the Nutrition Database System for Research (NDSR) 24-hour dietary recall. The NDSR is a dietary analysis software application used to collect and calculate nutritional intake.
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: grams
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
grams
  Baseline | 29.9 (3.5)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 32.2 (4.0)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 29.8 (4.4)

6. Secondary Outcome: Intake of Fruit
Description: The dietary behavior of consumption of fruit was measured by using the NDSR 24-hour dietary recall. The NDSR is a dietary analysis software application used to collect and calculate nutritional intake. The NDSR calculates the number of servings from 7 subcategories including citrus fruits, fruits other than citrus, avocado, as well as processed fruits. Serving amounts for all fruit are calculated by the NDSR software based on standard serving sizes for each specific food item. The total servings from all subcategories are reported here.
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: servings of fruit
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
servings of fruit
  Baseline | 2.2 (0.3)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 2.3 (0.5)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 1.7 (0.3)

7. Secondary Outcome: Intake of Vegetables
Description: The dietary behavior of consumption of vegetables was measured by using the NDSR 24-hour dietary recall. The NDSR is a dietary analysis software application used to collect and calculate nutritional intake. The NDSR calculates the number of servings from 10 subcategories including potatoes, juice, green or yellow vegetables, and legumes. Serving amounts for all fruit are calculated by the NDSR software based on standard serving sizes for each specific food item. The total servings from all subcategories are reported here.
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: servings of vegetables
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
servings of vegetables
  Baseline | 3.2 (0.3)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 3.7 (0.4)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 3.1 (0.3)

8. Secondary Outcome: Change in International Physical Activity Questionnaire (IPAQ) Score
Description: The International Physical Activity Questionnaire (IPAQ) includes 7-items asking respondents how many days in the past week they participated in vigorous, moderate and mild activities and how many minutes per day they spent on those activities. Data collected with IPAQ can be reported as a continuous measure and is computed by weighting each type of activity by its energy requirements defined in Metabolic Equivalent of Tasks (METs) to yield a score in MET-minutes (the MET score of an activity multiplied by the minutes performed). MET-minutes per week will be compared between study time points.
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: MET minutes per week
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
MET minutes per week
  Baseline | 2872.5 (613.8)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 4716.7 (683.4)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 5952.6 (1236.9)

9. Secondary Outcome: Waist Circumference
Description: Body composition will be assessed by waist circumference measured in centimeters (cm).
Time Frame: Baseline, Week 12, Week 24
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
Number analyzed (Participants) | 41
centimeters
  Baseline | 107.7 (1.6)
  Week 12: number analyzed (Participants) | 37
  Week 12 | 103.3 (1.5)
  Week 24: number analyzed (Participants) | 25
  Week 24 | 101.1 (1.5)

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected from the time participants began the intervention through the end of intervention assessment at Week 24.
Arm/Group | Soccer-based Adaptation to the Diabetes Prevention Program (DPP)
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 5/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soccer-based Adaptation to the Diabetes Prevention Program (DPP) (N=41)
Mild injuries (Musculoskeletal and connective tissue disorders) | 5 (5) — Hamstring strain, calf strain, or Achilles' tendinitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03595384/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03595384/ICF_001.pdf